CLINICAL TRIAL: NCT01349465
Title: A Prospective 3-Year Follow-up Study in Subjects Previously Treated in a Phase IIb or Phase III Study With a TMC435-Containing Regimen for the Treatment of Hepatitis C Virus (HCV) Infection
Brief Title: 3-year Follow-up Study in Patients Previously Treated With TMC435-Containing Regimen for the Treatment of Hepatitis C Virus Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR017365; TMC435HPC3002 (Other: Janssen R&D Ireland); 2010-019843-20 (EudraCT Number)
Record Dates: First submitted 2011-04-26; First posted 2011-05-06 (Estimated); Results first posted 2017-02-16 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Hepatitis; TMC435; Liver disease; Virus Infection
MeSH Terms: conditions — Hepatitis C; Hepatitis; Liver Diseases; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: TMC 435 - Patients With SVR at LPVPS (Other): Patients with sustained virologic response (SVR) who completed last post-therapy follow-up visit of the previous study (LPVPS) [Phase IIb or Phase III] in which they received a TMC435-containing regimen for the treatment of HCV infection.
  Interventions: Drug: No treatment
- Group 2: TMC 435 - Patients With No SVR at LPVPS (Other): Patients with no sustained virologic response (SVR) who completed last post-therapy follow-up visit of the previous study (LPVPS) [Phase IIb or Phase III] in which they received a TMC435-containing regimen for the treatment of HCV infection.
  Interventions: Drug: No treatment

INTERVENTIONS:
Drug: No treatment — No treatment was given to patients during this study as this is a follow-up study of previous Phase IIb or Phase III in which they received a TMC435-containing regimen.

SUMMARY:
The purpose of this study is to investigate durability of SVR in chronic HCV patients who achieved SVR in the previous study with TMC435-containing regimen and time for resistance associated mutations to return to baseline in chronic HCV patients who did not achieve SVR in the previous study with TMC435-containing regimen.

DETAILED DESCRIPTION:
This is a 3-year follow-up study in patients who completed the last post-therapy follow-up visit of the previous Phase IIb [NCT00882908, NCT00980330] or Phase III [NCT01289782, NCT01290679, NCT01281839] study in which they received TMC435, in combination with pegylated interferon and ribavirin, for the treatment of hepatitis C infection. The entire study duration for each patients will be approximately 36 months. The medical follow-up of the patients will be performed according to the local standard of care. This study will evaluate the levels of hepatitis C virus in the blood circulation, as well as safety and alpha-fetoprotein testing and the change in sequence of HCV NS3/4A region over time in patients with confirmed detectable HCV RNA at last post-therapy follow-up visit of the previous TMC435 study. In this study the development of liver disease progression will also be assessed. No medication will be administered in this study.

ELIGIBILITY:
Inclusion Criteria:

* Have previously participated in a Phase IIb or Phase III study
* Must have received at least one dose of TMC435 in that study
* Has completed the last post-therapy follow-up visit of the previous (LPVPS) study

Exclusion Criteria:

* Must be currently enrolled or plan to enroll in another study with an investigational drug or invasive investigational medical device
* Have received antiviral or immunomodulating treatment, including therapeutic vaccines, for hepatitis C virus (HCV) between LPVPS and the screening visit of present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2011-07-04 (Actual); Primary Completion 2016-01-05 (Actual); Study Completion 2016-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (48):
- United States (12):
  - Bakersfield, California
  - La Jolla, California
  - Los Angeles, California
  - Jacksonville, Florida
  - Orlando, Florida
  - Chicago, Illinois
  - New Orleans, Louisiana
  - Saint Paul, Minnesota
  - Tupelo, Mississippi
  - Chapel Hill, North Carolina
  - Cincinnati, Ohio
  - San Antonio, Texas
- Belgium (5):
  - Antwerp
  - Bruges
  - Brussels
  - Ghent
  - Leuven
- Canada (5):
  - Calgary, Alberta
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Montreal
- France (6):
  - Créteil
  - Grenoble
  - Lyon
  - Nice
  - Paris
  - Vandœuvre-lès-Nancy
- Germany (9):
  - Berlin
  - Cologne
  - Düsseldorf
  - Frankfurt A. M.
  - Freiburg im Breisgau
  - Hamburg
  - Hanover
  - Kiel
  - Würzburg
- Poland (5):
  - Bialystok
  - Bydgoszcz
  - Czeladź
  - Mysłowice
  - Warsaw
- Russia (6):
  - Moscow
  - Nizhny Novgorod
  - Saint Petersburg
  - Samara
  - Smolensk
  - Stavropol

REFERENCES:
- [Derived] Zoulim F, Moreno C, Lee SS, Buggisch P, Horban A, Lawitz E, Corbett C, Lenz O, Fevery B, Verbinnen T, Shukla U, Jessner W. A 3-year follow-up study after treatment with simeprevir in combination with pegylated interferon-alpha and ribavirin for chronic hepatitis C virus infection. Virol J. 2018 Jan 30;15(1):26. doi: 10.1186/s12985-018-0936-4. PMID 29378602

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total 250 participants were screened and among those 249 were enrolled into the study (200 participants with SVR and 49 participants with no SVR).
Groups:
- SVR at Last Post-Therapy Follow-up Visit of Previous Study: Participants with sustained virologic response (SVR) at last post-therapy follow-up visit of the previous Phase IIb [NCT00882908, NCT00980330] or Phase III [NCT01289782, NCT01290679, NCT01281839] study.
- No SVR at Last Post-Therapy Follow-up Visit of Previous Study: Participants with no sustained virologic response (SVR) at last post-therapy follow-up visit of the previous Phase IIb [NCT00882908, NCT00980330] or Phase III [NCT01289782, NCT01290679, NCT01281839] study.
Period: Overall Study
Arm/Group | SVR at Last Post-Therapy Follow-up Visit of Previous Study | No SVR at Last Post-Therapy Follow-up Visit of Previous Study
Started | 200 | 49
Completed | 182 | 27
Not Completed | 18 | 22
Not completed — Adverse Event | 1 | 0
Not completed — Death | 3 | 0
Not completed — Lost to Follow-up | 10 | 1
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Subject Ineligible To Continue The Trial | 0 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SVR at Last Post-Therapy Follow-up Visit of Previous Study | No SVR at Last Post-Therapy Follow-up Visit of Previous Study | Total
Number analyzed (Participants) | 200 | 49 | 249
Age, Continuous [Median (Full Range); unit: years] | 52 [22 to 70] | 56 [28 to 70] | 53 [22 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 17 | 95
  Male | 122 | 32 | 154

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Maintaining SVR at the Last Available Visit
Description: The SVR rate is the proportion (%) of participants with HCV RNA less than (<) 25 International Units/milliliter (IU/mL).
Time Frame: Last Available Visit (Month 36 for subjects completing the study)
Population: All participants with SVR at LPVPS were included in the population analysis set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SVR at Last Post-Therapy Follow-up Visit of Previous Study
Number analyzed (Participants) | 200
Percentage of participants | 100 [98.2 to 100]

2. Primary Outcome: Overall Percentage of Participants With Change in Sequence of HCV NS3/4A Region Over Time in Participants With Confirmed Detectable HCV RNA at the Last Visit of the Previous Study
Description: Sequencing was performed to assess changes in the sequence of the HCV NS3/4A protein region over time in participants with no SVR at LPVPS (ie confirmed detectable HCV RNA at the last visit of the previous study). EOS defined as last available sequencing sample. AEM and NEM represents any emerging mutation and no emerging mutation at time of failure of the previous study.
Time Frame: Baseline and Month 36
Population: "N" signifies number of participants with no SVR at LPVPS and with available sequence data. "n" defines the number of participants analyzed at specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | No SVR at Last Post-Therapy Follow-up Visit of Previous Study
Number analyzed (Participants) | 48
Percentage of participants
  NEM Return to Baseline at EOS (n=5) | 0.0 [46.7 to 230.3]
  NEM Change to New Profile at EOS (n=5) | 0.0
  AEM Return to Baseline at EOS (n=43) | 86.0
  AEM Change to New Profile at EOS (n=43) | 7.0

3. Secondary Outcome: Percentage of Participants With Late Viral Relapse
Description: Relapse at any time after the LPVPS until the last individual visit of this study. All participants maintained SVR until the last available visit. No late viral relapse was therefore observed.
Time Frame: End of study (at month 36)
Population: Late viral relapse was evaluated in all enrolled participants with SVR at LPVPS.
Measure: Number; unit: percentage of participants
Arm/Group | SVR at Last Post-Therapy Follow-up Visit of Previous Study
Number analyzed (Participants) | 200
percentage of participants | 0

4. Secondary Outcome: Number of Participants With Adverse Events (AEs) as a Measure of Safety and Tolerability
Time Frame: End of study (at month 36)
Measure: Number; unit: Participants
Arm/Group | SVR at Last Post-Therapy Follow-up Visit of Previous Study | No SVR at Last Post-Therapy Follow-up Visit of Previous Study
Number analyzed (Participants) | 200 | 49
Participants
  Adverse Events (AE) | 4 | 1
  Serious Adverse Events (SAE) | 10 | 0

5. Primary Outcome: Percentage of Participants With Change in Sequence of HCV NS3/4A Region Over Time in Participants With Confirmed Detectable HCV RNA (With Q80K at Baseline) at the Last Visit of the Previous Study
Description: as for outcome 2
Time Frame: Baseline and Month 36
Population: "N" signifies number of particpants with no SVR at LPVPS and with available sequence data. "n" defines the number of participants analyzed at specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | SVR at Last Post-Therapy Follow-up Visit of Previous Study
Number analyzed (Participants) | 10
Percentage of participants
  NEM Return to Baseline at EOS (n=1) | 0.0
  NEM Change to New Profile at EOS (n=1) | 0.0
  AEM Return to Baseline at EOS (n=9) | 88.9
  AEM Change to New Profile at EOS (n=9) | 0.0

6. Primary Outcome: Percentage of Participants With Change in Sequence of HCV NS3/4A Region Over Time in Participants With Confirmed Detectable HCV RNA (Without Q80K at Baseline) at the Last Visit of the Previous Study
Description: as for outcome 2
Time Frame: Baseline and Month 36
Population: as for outcome 5
Measure: Number; unit: Percentage of participnats
Arm/Group | SVR at Last Post-Therapy Follow-up Visit of Previous Study
Number analyzed (Participants) | 38
Percentage of participnats
  NEM Return to Baseline at EOS (n=4) | 0.0
  NEM Change to New Profile at EOS (n=4) | 0.0
  AEM Return to Baseline at EOS (n=34) | 85.3
  AEM Change to New Profile at EOS (n=34) | 8.8

ADVERSE EVENTS:
Time Frame: End of study (36 Months)
Description: Only Adverse Events associated with a study procedure or the use of any J&J medication were collected from signing of the Informed Consent Form onwards until the last study visit and classified according to the existing procedures. If during the study, hepatocellular carcinoma (HCC) was diagnosed, it should be reported as an AE.
Groups:
- Total: All Enrolled Subjects
Arm/Group | SVR at Last Post-Therapy Follow-up Visit of Previous Study | No SVR at Last Post-Therapy Follow-up Visit of Previous Study | Total
Serious Adverse Events (participants affected / at risk) | 10/200 | 0/49 | 10/249
Other Adverse Events (participants affected / at risk) | 4/200 | 1/49 | 5/249
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SVR at Last Post-Therapy Follow-up Visit of Previous Study (N=200) | No SVR at Last Post-Therapy Follow-up Visit of Previous Study (N=49) | Total (N=249)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 3
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 1 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 1
General physical health deterioration (General disorders) | 1 | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 1
Hydrocholecystis (Hepatobiliary disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SVR at Last Post-Therapy Follow-up Visit of Previous Study (N=200) | No SVR at Last Post-Therapy Follow-up Visit of Previous Study (N=49) | Total (N=249)
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Alpha 1 foetoprotein increased (Investigations) | 0 | 1 | 1
Dysarthria (Nervous system disorders) | 1 | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.